CLINICAL TRIAL: NCT06977282
Title: The 'Bone-Brain' Crosstalk Mechanism of Subchondral Bone Nociceptive Sensitization Activating SPP1-Positive Microglia in the vlPAG Region Elucidates the Theoretical Connotation of Treating Knee Osteoarthritis Based on Kidney Differentiation
Status: Not yet recruiting | Type: Observational
Sponsor: Jinchao Xu (Other)
Responsible Party: Sponsor-Investigator, Jinchao Xu, Resident Physician, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Other Study IDs: SPHFJP-S2025079-1
Record Dates: First submitted 2025-04-12; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tibial plateau samples obtained from KOA patients during total knee arthroplasty.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KOA: Patients with knee osteoarthritis of renal deficiency type who meet the diagnostic criteria
- HC: Healthy volunteers

SUMMARY:
The aim of this observational study is to investigate the relationship between pain severity and alterations in bone-derived and brain-derived signaling molecules (including serum neurotransmitters and inflammatory cytokines), as well as structural and functional changes in the ventrolateral periaqueductal gray (vlPAG) region in patients with kidney-deficiency type knee osteoarthritis (KOA). The central question it seeks to address is whether changes in these signaling molecules and vlPAG alterations are associated with the degree of pain.

Patients scheduled to undergo total knee arthroplasty (TKA) due to KOA will be enrolled prior to surgery. Before the operation, they will undergo questionnaire assessments, physical examinations, imaging evaluations, and blood sample collection. The resected tibial plateau tissue obtained during surgery will be used for subsequent laboratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of KOA
* Age between 60-70 years.
* Kellgren-Lawrence grade IV on anteroposterior and lateral knee X-rays.
* Scheduled for total knee arthroplasty.
* Voluntarily signs informed consent.

Exclusion Criteria:

* Clinical diagnosis of ankylosing spondylitis, rheumatoid arthritis, gout, or other related conditions.
* Presence of metabolic bone diseases, acute trauma, malignancies, infections, or other complications severely affecting knee function.
* Use of drugs affecting bone metabolism (e.g., corticosteroids, zoledronic acid) within the past 6 months.
* Presence of psychiatric disorders or serious cardiovascular, pulmonary, renal, hepatic, hematologic, or other systemic diseases.
* Contraindications to MRI.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis of kidney deficiency type from the Affiliated People's Hospital of Fujian University of Traditional Chinese Medicine. And the healthy volunteers recruited by the research team.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index | Participants were tested immediately after being included in the study.
  The WOMAC Index is a validated instrument used to assess pain, stiffness, and physical dysfunction in patients with osteoarthritis. It comprises 3 subscales with a total of 24 items, yielding a total score ranging from 0 to 96, where higher scores indicate more severe symptoms and greater functional impairment.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) score | Participants were tested immediately after being included in the study.
  The VAS score is a subjective measure used to assess pain intensity, typically presented as a continuous scale ranging from 0 to 10, with higher scores indicating greater pain severity.
Pattern Element Analysis | Participants were tested immediately after being included in the study.
  A pattern differentiation system would be used to assess the severity of kidney-deficiency-related pathological changes.
Function of Knee Joint | Participants were tested immediately after being included in the study.
  Gait analysis and neutral position (0°) method to evaluate knee joint function.
Volume of Subchondral Cystic Lesions | Participants were tested immediately after being included in the study.
  Knee MRI combined with Mimics software would be used to calculate the volume of subchondral cystic lesions.
Brain Region Structure | Participants were tested immediately after being included in the study.
  Diffusion Tensor Imaging (DTI) would be employed to investigate microstructural alterations in the vlPAG by assessing the diffusion properties of water molecules, thereby reflecting the integrity and connectivity of white matter tracts.
Brain Region Functional Connection | Participants were tested immediately after being included in the study.
  Resting-state functional magnetic resonance imaging (fMRI) would be used to investigate alterations in functional connectivity of the vlPAG.
Serum Neurotransmitters | Participants were tested immediately after being included in the study.
  Ultra-High Performance Liquid Chromatography-Tandem Mass Spectrometry (UHPLC-MS/MS) would be employed to detect changes in serum levels of excitatory and inhibitory neurotransmitters.
Serum Inflammatory Cytokines | Participants were tested immediately after being included in the study.
  Serum levels of inflammatory cytokines would be measured using the Luminex multiplex liquid-phase assay.
Microarchitecture of Subchondral Bone | One day following TKA surgery.
  Following TKA surgery, the resected tibial plateau would be collected for further analysis. Micro-computed tomography (micro-CT) would be employed to assess differences in subchondral bone microarchitecture between load-bearing and non-load-bearing regions
Morphological Differences of Cartilage and Subchondral | One month following TKA surgery.
  Hematoxylin and eosin (HE) staining would be used to examine the morphological differences in cartilage and subchondral bone between the load-bearing and non-load-bearing regions of the tibial plateau.
Subchondral Bone Osteoclast Activity | One month following TKA surgery.
  Tartrate-resistant acid phosphatase (TRAP) staining would be used to assess osteoclast activity in the subchondral bone of load-bearing and non-load-bearing regions.
Subchondral Bone Osteoblastic Activity | One month following TKA surgery.
  Alkaline phosphatase (ALP) staining would be used to assess osteoblastic activity in the subchondral bone of load-bearing and non-load-bearing regions.
Subchondral Bone Sensory Nerve Fiber Distribution | One month following TKA surgery.
  Karnovsky-Roots staining would be used to assess the distribution of sensory nerve fibers in the subchondral bone of load-bearing and non-load-bearing regions.
Pain-Sensitization-Related Factors in Subchondral Bone | One month following TKA surgery.
  Immunofluorescence staining would be used to evaluate changes in pain-sensitization-related regulatory factors in the subchondral bone (SPP1, Netrin1, TMEM119, PGE2, EP4) of load-bearing and non-load-bearing regions.
Subchondral Bone Osteoclast Marker | One month following TKA surgery.
  Immunofluorescence staining would be used to detect changes in osteoclast marker proteins (TRAP, CTSK) in the subchondral bone of load-bearing and non-load-bearing regions.
Subchondral Bone Nociceptor Distribution | One month following TKA surgery.
  Immunofluorescence staining would be used to detect changes in nociceptor marker proteins (TRPV1, TRPA1, CGRP, TrkA, NF200) in the subchondral bone of load-bearing and non-load-bearing regions.